CLINICAL TRIAL: NCT04141033
Title: Assessment of Salivary and Gingival Crevicular Fluid Neopterin Levels in Pre- and Post-menopausal Women With Chronic Periodontitis Following Nonsurgical Periodontal Therapy (A Clinical and Biochemical Study)
Brief Title: Assessment of Neopterin Levels in Pre- and Post-menopausal Women With Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Abeer Alaa El-Din, Master student at Ain Shams University Faculty of Dentistry, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Abeer Alaa 88
Record Dates: First submitted 2019-10-19; First posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Menopause
Keywords: Periodontitis; Neopterin; Menopausal women; Non-surgical periodontal therapy
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- saliva neopterin levels (Other): assessment of saliva neopterin levels in pre and post-menopausal women
  Interventions: Diagnostic Test: assessment of neopterin levels
- GCF neopterin levels (Other): assessment of GCF neopterin levels in pre and post-menopausal women
  Interventions: Diagnostic Test: assessment of neopterin levels

INTERVENTIONS:
Diagnostic Test: assessment of neopterin levels — neopterin is a macrophage biomarker used for diagnosis of active periodontitis and the response to treatment

SUMMARY:
Neopterin is an early and valuable biomarker of cellular immunity, shown to be a sensitive assessment parameter for cell-mediated immune reactions. Hence determination of neopterin concentrations in distinctive body fluids is of diagnostic interest in a wide range of T lymphocytes and macrophages originated diseases. Increased neopterin production is also found in infections due to intracellular living bacteria and parasites. Neopterin concentration is directly proportional to the reactive oxygen species levels and is inversely related to the serum concentration of antioxidants like alpha-tocopherol. Hence it can be regarded as a marker of reactive oxygen species formed by the activated cellular immune system. Consequentially this is useful for predicting the prognosis and diagnosis of severe form of periodontal diseases. Menopause accomplishes a wide range of changes in women's body, and the oral cavity is also not exceptional. As exalted levels of ovarian hormones, detected in pregnancy and oral contraceptive usage, can lead to an increase of gingival inflammation. On the contrary, menopause shows depleted levels of ovarian sex steroids, which also causes worsening of gingival health. Post-menopause was found to be more aggressive and destructive in nature compared to pre-menopause. It has been assessed that the prevalence of oral discomfort was found to be significantly higher along with low flow rates of the saliva with the presence of periodontal disease more frequently. Studies demonstrated that non-surgical periodontal therapy reduces inflammation and improves periodontal status. Therefore it can be assumed that overall inflammatory markers also reduce after non-surgical periodontal therapy.

DETAILED DESCRIPTION:
A total of 30 patients will be selected, 15 per-menopause and 15 post-menopausal women. Full mouth scaling and root planing will be performed. All clinical parameters will be recorded at the baseline visit before mechanical debridement and after 3 months of treatment. Saliva samples will be collected at the primary visit before scaling and root planing as a baseline value, and after 1 month and 3 months postoperatively. Gingival crevicular fluid (GCF) samples will be collected at the primary visit before scaling and root planing as a baseline value, and after 1 month and 3 months postoperatively. Neopterin will be measured in the samples using commercially available Enzyme Linked Immunosorbent Assay (ELISA) kit. Statistical analysis will be performed to the results.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged from (35- 60).
* Clinically diagnosed with chronic moderate periodontitis having more than 10 natural teeth and at least two teeth exhibiting clinical attachment loss (CAL) ≥4 mm.
* Systemically healthy individuals and not taking any hormonal therapy or drugs that affect hormonal status.
* Patient compliance

Exclusion Criteria:

* Smokers.
* Pregnant or lactating females.
* Periodontal treatment <6 months prior to the preliminary visit.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — subjects are categorized depending on menstrual history
Enrollment: 30 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
assess salivary and gingival crevicular fluid neopterin levels in patients with chronic periodontitis in pre- and post-menopausal women | 3 months
  measuring of neopterin levels using commercially available ELISA kit

SECONDARY OUTCOMES:
evaluate the value of neopterin as a biomarker | 3 months
  depending on the result, if neopterin is correleated with the disease activity it can be used as a biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Nevine H. Kheir El Din, Professor, Study Director — Faculty of Dentistry- Ain Shams University; Waleed M. Abbas, lecturer, Study Director — Faculty of Dentistry- Ain Shams University
Locations (1):
- Ain Shams University- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No